CLINICAL TRIAL: NCT07292675
Title: The Effect of Low Intensity Training With Blood Flow Restriction Versus Traditional Resistance Exercise on Lower Extermity Isokinetic Torque and Balance in Ischemic Stroke Patients
Brief Title: The Effect of Low Intensity With BFR on Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Ibrahim Ahmed Ibrahim Abu Ella, lecturer, Delta University for Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005961
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke
Keywords: BFR , Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Groups:
  * Group A: Low-intensity BFR resistance training
  * Group B: Traditional resistance training
Who Masked: Participant
Masking Description: The patients in control group will receive high intensity resistance training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Study group will receive low-intensity BFR resistance training
  Interventions: Other: low-intensity resistance training with blood flow restriction
- Control group (Active Comparator): Control group will receive high intensity resistance training
  Interventions: Other: High intensity resistance training

INTERVENTIONS:
Other: low-intensity resistance training with blood flow restriction — "Low-Intensity" BFR Means (for Quads)
  It involves resistance 20-30% 1RM combined with partial arterial + full venous restriction using a cuff placed on the proximal thigh.
  Arms: Study group
Other: High intensity resistance training — High-intensity quadriceps training in stroke patients focuses on using 60-80% of 1RM to improve strength, motor unit recruitment, and functional mobility. Exercises such as loaded sit-to-stand, leg press, and step-ups are commonly used to target the quadriceps safely. Training intensity is guided by a perceived exertion of 7-9/10 while maintaining proper supervision to prevent falls. This approach enhances knee stability, gait efficiency, and overall functional independence.
  Arms: Control group

SUMMARY:
To compare the effects of low-intensity resistance training with blood flow restriction (BFR) versus traditional resistance training on lower limb isokinetic torque and dynamic balance in ischemic stroke survivors.

DETAILED DESCRIPTION:
Ischemic stroke commonly results in reduced lower extremity muscle torque and impaired balance, affecting mobility and fall risk.

Traditional resistance training improves muscle function but may not be suitable for all patients due to the need for high mechanical loads.

Low-intensity resistance training with blood flow restriction (BFR) has emerged as an alternative that enhances muscular adaptation at lower loads. However, limited data exists on its effect on isokinetic torque and functional balance in stroke patients. This study aims to fill this gap using objective isokinetic measurements and validated balance scales.

ELIGIBILITY:
Inclusion Criteria:

* • First-ever ischemic stroke (3-12 months post-stroke)

  * Aged 30-40 years
  * Can walk independently or with an aid
  * Medically stable and able to follow instructions

Exclusion Criteria:

* •Hemorrhagic stroke

  * Deep vein thrombosis or peripheral vascular disease
  * Orthopedic conditions affecting lower limb
  * Severe cognitive impairment or uncontrolled hypertension

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-13 (Estimated); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-05-13 (Estimated)

PRIMARY OUTCOMES:
Isokinetic torque | Baseline

IPD SHARING:
Plan to Share IPD: No